CLINICAL TRIAL: NCT04958590
Title: The Standing and Sitting Spino-pelvic Sagittal Alignment in Chinese Population
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2018192
Record Dates: First submitted 2021-06-27; First posted 2021-07-12 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-06

CONDITIONS: Sagittal Alignment
Keywords: sagittal alignment; sitting; spinal fusion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1 （asymptomatic）: the middle-aged and elderly Chinese asymptomatic population who underwent the whole spine X-ray in standing and sitting positions.
  Interventions: Radiation: whole spine X-ray
- 2 （patients）: the patients who underwent posterior lumbar fusion surgery for lumbar degenerative disease has been followed up for three months.
  Interventions: Radiation: whole spine X-ray

INTERVENTIONS:
Radiation: whole spine X-ray — Group 1 underwent whole spine X-ray in standing and sitting positions.

SUMMARY:
This study is aimed to demonstrate the standing and sitting spino-pelvic sagittal alignment in Chinese population, then to explore the influence of spinal fusion on the changes when moving from standing to sitting positon.

ELIGIBILITY:
Inclusion Criteria:

Group 1 90 Healthy Volunteers - age >40 years, no history of neck pain, back pain, or radicular pain in the previous six months, no history of chronic neck or back pain lasting more than three months, no history of spinal disease or surgery, no spinal deformity or lumbar spondylolisthesis, no history of hip or knee arthroplasty or other realignment surgery of the lower extremities, and no history of neuromuscular disorders.

Group 2 126 patients Clinical diagnosis of Lumbar degenerative disease

Exclusion Criteria:

Group 1 90 Healthy Volunteers

- pregnant

Group 2 126 patients

* Neuromuscular diseases
* Arthritis
* Tumor
* A previous history of lumbar fusion surgery

Ages: 42 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Volunteers Patients with lumbar degenerative disease who had undergone surgery in Peking university third hospital.
Sampling Method: Non-Probability Sample
Enrollment: 216 (Actual)
Dates: Start 2019-02-20 (Actual); Primary Completion 2019-09-09 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Group 2 The sagittal spinal parameters in degrees | 3 months after surgery
  The parameters included TPA (T1 pelvic angle,the angle between the line from the axis of the femoral head to the center of T1 and the line from the axis of the femoral head to the midpoint of the S1 endplate), lumbar lordosis (LL,the angle between the upper endplate of L1 and S1), thoracic kyphosis (TK,The angle between the upper endplate of T4 and the lower endplate of T12), pelvic incidence (PI,The angle between the line perpendicular to the midpoint of the sacral plate and the line connecting this to the midpoint of the hip axis), pelvic tilt (PT,The angle between the line from the middle of the sacral plate to the middle of the hip axis and the vertical line), sacral slope (SS,The angle between the sacral endplate and the horizontal line)
Group 1 The sagittal spinal parameters in degrees | 6 months after study started
  The parameters included TPA (T1 pelvic angle,the angle between the line from the axis of the femoral head to the center of T1 and the line from the axis of the femoral head to the midpoint of the S1 endplate), lumbar lordosis (LL,the angle between the upper endplate of L1 and S1), thoracic kyphosis (TK,The angle between the upper endplate of T4 and the lower endplate of T12), pelvic incidence (PI,The angle between the line perpendicular to the midpoint of the sacral plate and the line connecting this to the midpoint of the hip axis), pelvic tilt (PT,The angle between the line from the middle of the sacral plate to the middle of the hip axis and the vertical line), sacral slope (SS,The angle between the sacral endplate and the horizontal line)
Group 1 The sagittal spinal parameters in millimeter | 6 months after study started
  SVA (sagittal vertical axis, The offset between the center of C7 and the plumb line drawn from posterosuperior corner of S1)

SECONDARY OUTCOMES:
Group 2 Disability assessed by the Oswestry Disability Index (ODI) | 3 months after surgery
  The Oswestry Disability Index (ODI) (0-100) is used to assess disability.Higher scores mean a worse outcome.
Group 2 Back pain assessed by the VAS | 3 months after surgery
  The Visual Analog Scale (0-10) is used to evaluate back pain.Higher scores mean a worse outcome
Group 2 Leg pain assessed by the VAS | 3 months after surgery
  The Visual Analog Scale (0-10) is used to evaluate leg pain.Higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Shi Li, Dr., Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Lafage R, Schwab F, Challier V, Henry JK, Gum J, Smith J, Hostin R, Shaffrey C, Kim HJ, Ames C, Scheer J, Klineberg E, Bess S, Burton D, Lafage V; International Spine Study Group. Defining Spino-Pelvic Alignment Thresholds: Should Operative Goals in Adult Spinal Deformity Surgery Account for Age? Spine (Phila Pa 1976). 2016 Jan;41(1):62-8. doi: 10.1097/BRS.0000000000001171. PMID 26689395
- [Background] Hey HWD, Teo AQA, Tan KA, Ng LWN, Lau LL, Liu KG, Wong HK. How the spine differs in standing and in sitting-important considerations for correction of spinal deformity. Spine J. 2017 Jun;17(6):799-806. doi: 10.1016/j.spinee.2016.03.056. Epub 2016 Apr 7. PMID 27063999
- [Background] Cho KJ, Suk SI, Park SR, Kim JH, Kang SB, Kim HS, Oh SJ. Risk factors of sagittal decompensation after long posterior instrumentation and fusion for degenerative lumbar scoliosis. Spine (Phila Pa 1976). 2010 Aug 1;35(17):1595-601. doi: 10.1097/BRS.0b013e3181bdad89. PMID 20386505